CLINICAL TRIAL: NCT04728087
Title: ACCEL® Absorbable Hemostat Powder Clinical Trial
Brief Title: ACCEL Absorbable Hemostat
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hemostasis, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Protocol 0312
Record Dates: First submitted 2021-01-21; First posted 2021-01-28 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2023-11

CONDITIONS: Hemostasis
MeSH Terms: interventions — Gelatin Sponge, Absorbable

STUDY DESIGN:
Who Masked: Participant
Masking Description: Sealed, blinded envelopes will be provided by the Sponsor (Hemostasis LLC). The Investigator/designee only opens the randomization envelope after the subject has been deemed eligible for the study and an eligible TBS has been identified in order to reduce potential bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- ACCEL (Experimental): Participant will be treated with up to 2 bellows (10 grams nominal) of ACCEL®.
  Interventions: Device: ACCEL® Absorbable Hemostat Powder
- Gelfoam or SURGIFOAM (Active Comparator): Participant will be treated with up to 12.5 cm x 8.0 cm of Gelfoam® (Absorbable Gelatin Sponge, Pfizer Manufacturer Part Number 0342-01) or SURGIFOAM® (Absorbable Gelatin Sponge, Manufacturer Part Number ETH1974).
  Interventions: Device: Gelfoam® (Absorbable Gelatin Sponge, Pfizer Manufacturer Part Number 0342-01)

INTERVENTIONS:
Device: ACCEL® Absorbable Hemostat Powder — Up to 2 bellows (10 grams nominal) of ACCEL®
  Arms: ACCEL
Device: Gelfoam® (Absorbable Gelatin Sponge, Pfizer Manufacturer Part Number 0342-01) — Up to 12.5 cm x 8.0 cm of Gelfoam® or SURGIFOAM® .
  Other Names: SURGIFOAM® (Absorbable Gelatin Sponge, Manufacturer Part Number ETH1974).
  Arms: Gelfoam or SURGIFOAM

SUMMARY:
The ACCEL® Absorbable Hemostat Powder Clinical IDE Trial is designed as a prospective, multi-center, randomized, non-inferiority, controlled pivotal clinical trial to evaluate the safety and efficacy of the ACCEL® Absorbable Hemostat Powder as compared to gelatin sponge, for achieving hemostasis in subjects undergoing cardiovascular, liver, or soft tissue surgery, when control of oozing to moderate bleeding by standard surgical techniques is ineffective and/or impractical.

ELIGIBILITY:
Inclusion Criteria:

Pre-Surgery:

1. Subject is greater than or equal to 22 years old
2. Subject is undergoing a cardiovascular surgery, liver surgery or soft tissue surgical procedure
3. Subject is willing and able to provide appropriate (Institutional Review Board (IRB) approved) informed consent.
4. The subject is willing and able to comply with the requirements of the protocol, including follow-up evaluations and schedule.
5. The subject is willing to be treated with ACCEL® Absorbable Hemostat Powder
6. The subject is willing to be treated with a commercially available absorbable gelatin sponge

   During Surgery:
7. Subject has not received blood transfusions between screening and application of investigational product or commercially available absorbable gelatin sponge
8. There is an estimated TBS surface area of ≤ 60 cm2
9. Visual observation of oozing (0.01 g/10s ˂ Flow ˂ 0.04 g/10s), mild (0.04 g/10s ≤ Flow ˂ 0.32 g/10s), or moderate (0.32 g/10s ≤ Flow ˂ 1.01 g/10s) bleeding as validated and when control by conventional surgical techniques, including but not limited to suture, ligature and cautery, is ineffective and/or impractical
10. There is an absence of intra-operative complications other than bleeding, which, in the opinion of the Investigator, may interfere with the assessment of efficacy or safety
11. There has been no intra-operative use of adjunct hemostat(s) on the target bleeding site identified for application of the study treatment

Exclusion Criteria:

Pre-Surgery:

1. The subject is pregnant (verified in a manner consistent with institution's standard of care)
2. Subject is lactating
3. Subject is currently participating in another investigational device or drug trial or has participated in one in the past 4 weeks (prior to surgery) or is planning to participate in another research study involving any investigational product within 4 weeks after surgery
4. Subject is a prisoner, a minor or unable to adequately give informed consent due to mental or physical condition
5. Subject has medical, social, or psychosocial issues that the Investigator believes could impact the subject's safety or compliance with study procedures
6. Subject has a known allergy to potatoes
7. Subject has a known allergy to porcine collagen/gelatin
8. Subject has a religious or other objection to porcine products
9. Subject is unwilling to receive blood products
10. Subject has history of heparin-induced thrombocytopenia (only for cardiovascular subjects where heparin use is required)
11. Subject with a baseline abnormality of INR > 2.5 or an aPTT> 100 seconds during screening that is not explained by current drug treatment (e.g. heparin, warfarin, etc.).
12. Subjects with platelets < 100 X 109 PLT/L during screening
13. Subject with Aspartate Aminotransferase (AST) or Alanine aminotransferase (ALT) > 3 X upper limit normal range during screening, except for subjects undergoing liver resection surgery or with a diagnosis of liver metastases where there is no upper limit normal for these analytes due to the nature of their disease
14. Subject is unwilling or unable to return for the required follow-up after surgery

    During Surgery:
15. Subject has an operative bleeding site which the surgeon is unable or unwilling to control with a hemostatic agent
16. Extracorporeal cardiopulmonary bypass circuits or blood salvage circuits are to be used during or after identification of the TBS.
17. There has been intra-operative use of thrombin on the patient.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2021-10-26 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Demonstration of non-inferiority | Day 0 / Surgery
  Comparison of the percentage of subjects achieving hemostasis within three (3) minutes for cardiovascular surgery and within five (5) minutes for liver surgery and soft tissue surgery of the TBS using the ACCEL® Absorbable Hemostat Powder as compared to the control hemostat.
Determination of incidence of SADE and ADE | Through the six (6) week follow-up.
  The analysis and comparison of the incidence of SADEs and ADEs through the six (6) week follow-up endpoint for the ACCEL® Absorbable Hemostat Powder and the control hemostat.

SECONDARY OUTCOMES:
Determination of TTH | Day 0 / Surgery
  A comparison of TTH (either 90 seconds or 3 minutes for cardiovascular and either 2 minutes or 5 minutes for liver surgery and soft tissue surgery) for the application of ACCEL® Absorbable Hemostat Powder and the control hemostat on the TBS.
Individual subject success rate | Through the six (6) week follow-up.
  A comparison of the proportion of individual subject successes (i.e., successful hemostasis and no SADEs and ADEs) for the application of ACCEL® Absorbable Hemostat Powder and the control hemostat on the TBS.
Length of individual subject hospitalization | Through the post-surgical follow-up (Day 1-7)
  The calculation and comparison of the number of days of individual subject hospitalization through the post-surgical (Day 1-7) follow-up endpoint for the ACCEL® Absorbable Hemostat Powder and the control hemostat.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Keck Medical Center of USC, Los Angeles, California
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Washington University in St. Louis, St Louis, Missouri
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Wisconsin - Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No